CLINICAL TRIAL: NCT04391023
Title: The Effects of 2 mA and 4 mA Cerebellar Transcranial Direct Current Stimulation and Balance Training to Reduce Fall Risk in People With Multiple Sclerosis
Brief Title: Cerebellar tDCS and Balance Training in PwMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Alexandra Fietsmam, PhD Student, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201912430
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Brain Stimulation; Balance Training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Sham tDCS (Sham Comparator): The tDCS device will perform a 30 second ramp up to 2 mA and then an immediate 30 second ramp down to 0 mA. Until the 19:30 minute time point, the tDCS will remain at 0 mA. At this time point, the tDCS will ramp up to 2 mA and then will immediately ramp back down to 0 mA.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS); Behavioral: Balance Training
- 2 mA tDCS (Experimental): The participants in this group will receive tDCS at 2 mA while seated comfortably. The intensity will start at 0 mA and will be incrementally increased to the target intensity (2 mA) over the initial 30 seconds. Then, the tDCS will deliver stimulation at the target intensity until the 19:30 minute time point. At this point, the current will gradually decrease back to 0 mA.
  Interventions: Behavioral: Balance Training; Device: 2 mA Transcranial Direct Current Stimulation
- 4 mA tDCS (Experimental): The participants in this group will receive tDCS at 4 mA while seated comfortably. The intensity will start at 0 mA and will be incrementally increased to the target intensity (4 mA) over the initial 30 seconds. Then, the tDCS will deliver stimulation at the target intensity until the 19:30 minute time point. At this point, the current will gradually decrease back to 0 mA.
  Interventions: Behavioral: Balance Training; Device: 4 mA Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Sham Transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive brain stimulation technique in which a very weak electrical current (2 mA) is applied to the scalp at the beginning of the session and then remains at 0 mA for the duration of the session to control for placebo-like effects. The anode and cathode will both be placed over the cerebellum.
  Other Names: tDCS
  Arms: Sham tDCS
Behavioral: Balance Training — The balance training protocol will include balance training exercises on both compliant (i.e., foam pad and trampoline) and firm surfaces.
Device: 2 mA Transcranial Direct Current Stimulation — tDCS is a non-invasive brain stimulation technique in which very weak electrical current (2 mA) is applied to the scalp for 20 minutes. The anode and cathode will both be placed over the cerebellum.
  Other Names: tDCS
  Arms: 2 mA tDCS
Device: 4 mA Transcranial Direct Current Stimulation — tDCS is a non-invasive brain stimulation technique in which very weak electrical current (4 mA) is applied to the scalp for 20 minutes. The anode and cathode will both be placed over the cerebellum.
  Other Names: tDCS
  Arms: 4 mA tDCS

SUMMARY:
Many people with multiple sclerosis (PwMS) have decreased balance and postural control, gait deficits, and a high frequency of falls. High fall rates and mobility impairments pose a significant risk to the independence and quality of life of PwMS. Therefore, effective interventions to improve balance and postural control are urgently needed to decrease the frequency of falls in PwMS. Balance training has been demonstrated to significantly improve postural control and gait in PwMS. One possible treatment modality to amplify the effects of balance training is transcranial direct current stimulation (tDCS), a non-invasive means to increase cortical excitability and potentially prime the brain for task specific learning. The cerebellum plays a vital role in balance and posture and may be an important target structure for tDCS studies seeking to reduce fall risk. Studies have shown that anodal cerebellar tDCS is effective in improving balance control in older adults with high fall risk and patients with chronic stroke. However, the most effective tDCS intensity and the duration of the effects on balance control has not been established. Moreover, no study has combined cerebellar tDCS and balance training to reduce fall risk in PwMS. The purpose of this study is to investigate the effects of cerebellar transcranial direct current stimulation (tDCS) on fall risk in people with relapsing-remitting multiple sclerosis. We will conduct tDCS or SHAM followed by balance training on 4 consecutive days. We will evaluate fall risk with well-established functional tasks, such as the Berg Balance Scale, Timed Up and Go (TUG), the six minute walk test (6MWT), and static posturography.

Prospective participants, men and women with relapsing-remitting MS, will be recruited. To accomplish this study, 30 participants will be randomly assigned into 3 groups (2 mA tDCS, 4 mA tDCS, or SHAM). This study involves 4 daily visits at the Integrative Neurophysiology Lab at the same time of day for each subject and three follow-up visits. The duration of visit 1 will be approximately 2.5 hours and the duration of visits 2-4 will be approximately 1.5 hours. Visit 5, 6, and 7 will be approximately 24 hours, 1 week, and 3 weeks, respectively, after visit 4 and will last approximately 1.5 hours. During tDCS sessions, participants will undergo either Sham, 2 mA, and 4 mA tDCS for 20 minutes followed by balance training.

ELIGIBILITY:
Inclusion Criteria:

1. medically diagnosed with relapsing-remitting multiple sclerosis
2. 18-70 years of age
3. moderate disability (score of 2-6 on the Patient Determined Disease Scale)
4. self-reported differences in function between legs, have fallen within the last year
5. able to walk for 6 mins, and not taking any psychoactive medication.

Exclusion Criteria:

1. relapse within the last 60 days
2. have changed disease modifying medications in the last 45 days
3. are currently pregnant
4. have a concurrent neurological or neuromuscular disease
5. have been hospitalized within the last 90 days
6. have any contraindications for the tDCS device (i.e., pacemakers or metal implants)
7. are unable to understand/sign the consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Fietsam, M.S., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were assigned to the 2 mA tDCS group
Period: Overall Study
Arm/Group | Sham tDCS | 4 mA tDCS
Started | 9 | 9
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS | 4 mA tDCS | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.57 (11.04) | 50.57 (14.89) | 50.57 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Fatigue Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The FSS consists of nine statements used to assess perceived fatigability. Subjects are asked to rate how much they felt a statement applied to them, on a 7-point scale (low value = does not apply, high value = high agreement with the statement). The questionnaire is scored by calculating the average response to the statements. Therefore, the scores will range from 1 to 7 (1 = low fatigue, 7 = high fatigue). A score ≥ 4 indicates a clinically significant level of fatigue.
  units on a scale | 4.48 (1.68) | 3.14 (1.36) | 4.17 (1.50)
Functional Gait Assessment [Mean (Standard Deviation); unit: units on a scale] — The Functional Gait Assessment (FGA) assess postural stability and the ability of the subjects to perform motor tasks during walking. These tasks include demonstrating a change in gait speed, head turns during walking, and walking with a narrow base of support. The assessment consists of 10 tasks that are rated by an administrator on scale from 0 (severe impairment) to 3 (normal). Therefore, scores range from 0-30, with 30 being the highest score possible (normal ambulation).
  units on a scale | 24.71 (4.86) | 23.14 (9.04) | 23.93 (6.77)
Berg Balance Scale [Mean (Standard Deviation); unit: units on a scale] — The Berg Balance Scale (BBS) is a valid and reliable assessment of balance during static (e.g., standing with eyes closed) and dynamic conditions (e.g., completing a 360-degree turn) conditions. BBS scores range from 0 to 56. Lower scores indicate increased impairment in balance. A cut-off score of 44 has been established as a criterion to identify people with MS with a high fall risk.
  units on a scale | 53 (4.93) | 50 (11.56) | 51.73 (8.41)
Six Minute Walk Test [Mean (Standard Deviation); unit: meters] | 431.51 (86.09) | 481.30 (35.73) | 460.72 (70.40)
Timed Up and Go [Mean (Standard Deviation); unit: seconds] | 8.15 (1.55) | 8.78 (3.54) | 8.42 (2.55)

OUTCOME MEASURES:

1. Primary Outcome: Score on the Berg Balance Scale
Description: The BBS is a valid and reliable assessment of balance during static (e.g., standing with eyes closed) and dynamic conditions (e.g., completing a 360-degree turn) conditions. BBS scores range from 0 to 56. Lower scores indicate increased impairment in balance. A cut-off score of 44 has been established as a criterion to identify PwMS with a high fall risk.
Time Frame: 24 hours, 2 weeks, and 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS | 4 mA tDCS
Number analyzed (Participants) | 7 | 7
units on a scale
  24 hours post-intervention | 54.43 (2.37) | 51.43 (9.11)
  2-weeks post-intervention | 54.67 (2.07) | 50.33 (10.21)
  4-weeks post-intervention | 54.29 (2.56) | 51.17 (9.93)

2. Primary Outcome: Time to Complete the Timed Up and Go Test (TUG)
Description: The TUG measures the time it takes for the participant to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. Two trials were completed and the reported score is the average time between the two trials. A higher number means it took the participant more time to complete the task (i.e., worse performance).
Time Frame: 24 hours, 2 weeks, and 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sham tDCS | 4 mA tDCS
Number analyzed (Participants) | 7 | 7
seconds
  24 hours post-intervention | 7.81 (1.66) | 7.47 (3.78)
  2-week post-intervention | 7.55 (1.43) | 6.99 (3.34)
  4-weeks post-intervention | 7.10 (1.23) | 6.88 (3.10)

3. Secondary Outcome: Time to Complete the Six Minute Walk Test (6MWT)
Description: Subjects performed the 6MWT in a cordoned-off hallway with two symbols on the ground, placed 30 meters apart. Subjects were instructed to walk as far as possible between the marks for 6 minutes, walking around each symbol like a cone. Higher scores indicate more distance walked (i.e., better performance).
Time Frame: 24 hours, 2 weeks, and 4 weeks post-intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sham tDCS | 4 mA tDCS
Number analyzed (Participants) | 7 | 7
meters
  24 hours post-intervention | 464.04 (107.68) | 523.31 (44.70)
  2-weeks post-intervention | 479.33 (137.44) | 542.15 (91.86)
  4-weeks post-intervention | 487.44 (114.10) | 545.03 (104.95)

4. Secondary Outcome: Score on the Fatigue Severity Scale (FSS)
Description: The FSS consists of nine statements used to assess perceived fatigability. Subjects are asked to rate how much they felt a statement applied to them, on a 7-point scale (low value = does not apply, high value = high agreement with the statement). The questionnaire is scored by calculating the average response to the statements. Therefore, the scores will range from 1 to 7 (1 = low fatigue, 7 = high fatigue). A score ≥ 4 indicates a clinically significant level of fatigue.
Time Frame: 24 hours, 2-weeks, and 4-weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS | 4 mA tDCS
Number analyzed (Participants) | 7 | 7
units on a scale
  24 hours post-intervention | 4.21 (1.38) | 3.62 (2.11)
  2-weeks post-intervention | 3.81 (1.52) | 4.39 (1.31)
  4-weeks post-intervention | 3.60 (1.51) | 3.80 (1.64)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through follow-up with each participating. This was from the familiarization session to the 4-week follow-up (~6-weeks total).
Arm/Group | Sham tDCS | 4 mA tDCS
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04391023/Prot_SAP_000.pdf